CLINICAL TRIAL: NCT04627623
Title: Prevalence and Risk Factors of COVID-19 Infection in the Upper Silesian Agglomeration Population in 2020
Brief Title: Prevalence and Risk Factors of COVID-19 in the Upper Silesian Agglomeration
Acronym: EpiSARS2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Prof. Grzegorz Brożek, MD PhD, Prof. Grzegorz Brożek, MD PhD, Medical University of Silesia
Other Study IDs: 2020/ABM /COVID19/0044
Record Dates: First submitted 2020-11-12; First posted 2020-11-13 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Covid19; Respiratory Tract Infections; Severe Acute Respiratory Syndrome; Corona Virus Infection; RNA Virus Infections; Virus Disease; Respiratory Tract Disease
Keywords: Covid19; Risk factors; Prevalence; Mortality; anti-SARS-CoV-2 antibodies
MeSH Terms: conditions — COVID-19; Respiratory Tract Infections; Severe Acute Respiratory Syndrome; Coronavirus Infections; RNA Virus Infections; Virus Diseases; Respiratory Tract Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 5 ml venous blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screened arm: 6000 peoples (3x2000) in all ages randomly selected from the general population of three towns (Katowice, Sosnowiec, Gliwice).
  From all invited is collected a venous blood samples (5ml) to assay IgM and IgG antibodies.
  Interventions: Diagnostic Test: IgM and IgG antibodies assay

INTERVENTIONS:
Diagnostic Test: IgM and IgG antibodies assay — 5 ml venous blood sample collection to assay IgM and IgM against COVID19

SUMMARY:
Project is designed as a comprehensive population-based epidemiological study in Upper-Silesian Conurbation (Poland) aiming at:

1. analysis of available data on incidence and mortality due to COVID-19 and
2. estimation of the occurrence of viral infection SARS-CoV-2 as revealed by the results of serological test (ELISA: IgM, IgG), with assessment of risk factors.

The project's objectives are: to assess incidence and mortality due COVID-19 according to sex, age and coexisting diseases; to determine the level of potential "underdiagnosis" of the magnitude of COVID-19 mortality using vital statistics data for Upper-Silesian Conurbation; to assess the prevalence of SARS-CoV-2 based on the level of seropositivity in Upper-Silesian Conurbation; to identify host-related and environmental risk factors if the infection. Analysis of existing data will include monthly records on incidence and mortality over the period 01.01.2020-31.12.2020 and comparison of the findings with the monthly records of 2018 and 2019, for the same population. Cross-sectional epidemiological study will be located in three towne (Katowice, Sosnowiec, Gliwice). In each town a representative age-stratified sample of 2000 subjects will undergo questionnaire assessment and serological examination performed by serological test. The project corresponds with analogous population-based studies on COVID-19 in a number of countries and responds to the WHO recommendation in that field.

DETAILED DESCRIPTION:
Project is designed as a comprehensive population-based epidemiological study in Upper-Silesian Conurbation (Poland) aiming at:

1. analysis of available data on incidence and mortality due to COVID-19 and
2. estimation of the occurrence of viral infection SARS-CoV-2 as revealed by the results of serological test (ELISA: IgM, IgG), with assessment of risk factors.

The project's objectives are: to assess incidence and mortality due COVID-19 according to sex, age and coexisting diseases; to determine the level of potential "underdiagnosis" of the magnitude of COVID-19 mortality using vital statistics data for Upper-Silesian Conurbation; to assess the prevalence of SARS-CoV-2 based on the level of seropositivity in Upper-Silesian Conurbation; to identify host-related and environmental risk factors if the infection. Analysis of existing data will include monthly records on incidence and mortality over the period 01.01.2020-31.12.2020 and comparison of the findings with the monthly records of 2018 and 2019, for the same population. Cross-sectional epidemiological study will be located in three towne (Katowice, Sosnowiec, Gliwice). In each town a representative age-stratified sample of 2000 subjects will undergo questionnaire assessment and serological examination performed by serological test. The project corresponds with analogous population-based studies on COVID-19 in a number of countries and responds to the WHO recommendation in that field.

ELIGIBILITY:
Inclusion Criteria: citizens of one of three towns (Katowice, Sosnowiec, Gliwice) with no age limits

Exclusion Criteria: person who is not able to contact laboratory and obtain blood sample.

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Selected by random inhabitants of one of three towns (Katowice, Sosnowiec, Gliwice) with no age limits.
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2020-06-22 (Actual); Primary Completion 2021-03-22 (Estimated); Study Completion 2021-04-22 (Estimated)

PRIMARY OUTCOMES:
Estimation of prevalence of specific anti-SARS-CoV-2 IgM and IgG antibodies in general population. | 8 months
  Estimation of real prevalence of elevated IgM and IgG COVID antibodies in general population will allow to estimate real number of current and past COVID infection in the population.

SECONDARY OUTCOMES:
Frequency of asymptomatic course of COVID in individuals with anti-SARS-CoV2 antibodies | 8 months
  Prevalence of asymptomatic cases into seropositive population

CONTACTS AND LOCATIONS:
Overall Officials: Jan E Zejda, Prof, Principal Investigator — Medical University of Silesia in Katowice Poland
Locations (1):
- Diagnostyka sp zoo, Katowice, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pan Y, Li X, Yang G, Fan J, Tang Y, Zhao J, Long X, Guo S, Zhao Z, Liu Y, Hu H, Xue H, Li Y. Serological immunochromatographic approach in diagnosis with SARS-CoV-2 infected COVID-19 patients. J Infect. 2020 Jul;81(1):e28-e32. doi: 10.1016/j.jinf.2020.03.051. Epub 2020 Apr 10. PMID 32283141
- [Background] Li Z, Yi Y, Luo X, Xiong N, Liu Y, Li S, Sun R, Wang Y, Hu B, Chen W, Zhang Y, Wang J, Huang B, Lin Y, Yang J, Cai W, Wang X, Cheng J, Chen Z, Sun K, Pan W, Zhan Z, Chen L, Ye F. Development and clinical application of a rapid IgM-IgG combined antibody test for SARS-CoV-2 infection diagnosis. J Med Virol. 2020 Sep;92(9):1518-1524. doi: 10.1002/jmv.25727. Epub 2020 Apr 13. PMID 32104917
- [Background] Zhao J, Yuan Q, Wang H, Liu W, Liao X, Su Y, Wang X, Yuan J, Li T, Li J, Qian S, Hong C, Wang F, Liu Y, Wang Z, He Q, Li Z, He B, Zhang T, Fu Y, Ge S, Liu L, Zhang J, Xia N, Zhang Z. Antibody Responses to SARS-CoV-2 in Patients With Novel Coronavirus Disease 2019. Clin Infect Dis. 2020 Nov 19;71(16):2027-2034. doi: 10.1093/cid/ciaa344. PMID 32221519
- [Background] Lee CY, Lin RTP, Renia L, Ng LFP. Serological Approaches for COVID-19: Epidemiologic Perspective on Surveillance and Control. Front Immunol. 2020 Apr 24;11:879. doi: 10.3389/fimmu.2020.00879. eCollection 2020. PMID 32391022